CLINICAL TRIAL: NCT07071701
Title: A Clinical Trial to Observe the Safety of 23-Valent Pneumococcal Polysaccharide Vaccine in Target Population Aged 2 Years and Above
Brief Title: A Clinical Trial to Observe the Safety of 23-Valent Pneumococcal Polysaccharide Vaccine in Target Population
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-PPV-MA4002-JS
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acitive safety surveillance group
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: Influenza vaccine
- Passive safety surveillance group
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine; Biological: Influenza vaccine

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — 23-valent pneumococcal polysaccharide vaccine
Biological: Influenza vaccine — Influenza vaccine

SUMMARY:
An open clinical trial of a 23-valent pneumococcal polysaccharide vaccine (PPV23) developed by Sinovac Life Science Co., Ltd was conducted to evaluate the safety of Sinovac PPV23 in target population of individuals aged 2 years and above. All participants received 1 dose of PPV23 and self-selected whether to receive 1 dose of influenza vaccine at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily and at their own expense received the 23-valent pneumococcal polysaccharide vaccine;
* Participants and/or their guardians are able to understand and voluntarily participate in this study and sign an informed consent form;
* Provide valid legal identification.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged 2 years old and above.
Sampling Method: Non-Probability Sample
Enrollment: 19267 (Actual)
Dates: Start 2022-07-02 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions to 23-valent pneumonia vaccine within 0-28 days after single and combined vaccination. | 28 days after the vaccination

SECONDARY OUTCOMES:
Incidence of adverse events to 23-valent pneumonia vaccine within 0-28 days after single and combined vaccination. | 28 days after the vaccination
Incidence of adverse events to 23-valent pneumonia vaccine within 0-7 days after single and combined vaccination. | 7 days after the vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease Prevention and Control, Nanjing, Jiangsu, China